CLINICAL TRIAL: NCT00565045
Title: Contralaterally Controlled Functional Electrical Stimulation for Hemiparetic Hand
Brief Title: Treatments for Recovery of Hand Function in Acute Stroke Survivors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Case Western Reserve University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jayme Knutson, Assistant Professor, Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21HD054749 (NIH)
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Stroke, Acute; Stroke; Hemiparesis; Hemiplegia
Keywords: hand; stroke; hemiplegia; electrical stimulation; recovery
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCFES (Experimental): CCFES - Contralaterally Controlled Functional Electrical Stimulation
  * Stimulation to finger and thumb extensors and flexors only in response to and with an intensity proportional to opening and closing of the contralateral unimpaired hand
  * A glove instrumented with sensors and worn on the unimpaired hand detects the degree of hand opening and determines stimulation intensity
  * Therapy sessions are done with the subject being assisted by the CCFES system.
  Interventions: Device: Neuromuscular electrical stimulator
- cNMES (Active Comparator): cNMES - Cyclic NeuroMuscular Electrical Stimulation.
  * Preprogrammed cycles of finger and thumb flexor and extensor stimulation repeatedly and automatically close and open the hand without any effort or voluntary intent required by the subject.
  * Subject instructed to relax, not attempt to assist the stimulation, and not to move the contralateral arm/hand during stimulation
  * Therapy sessions are done without the stimulation system
  Interventions: Device: Neuromuscular electrical stimulator

INTERVENTIONS:
Device: Neuromuscular electrical stimulator — Intervention Characteristics Common to Both Groups
  • 6-week intervention
  1. Home "exercise", daily
     1. Exercise (at home) 2 sessions/day
     2. A "session" consists of 3 (for CCFES) or 4 (for cNMES) 15-min sets separated by 5 min rest
     3. A "set" entails hand opening, closing, and relaxing in response or synchrony to light and sound cues and according to group-specific instructions
  2. Lab "therapy", 2x/week
     1. Two 1.5-hr sessions/week, working on functional hand tasks and tracking task (if possible).

SUMMARY:
Impaired hand function is one of the most frequently persisting consequences of stroke. The purpose of this study is to investigate whether two different types of treatment improve recovery of hand function after stroke.

DETAILED DESCRIPTION:
Loss of hand function is common after stroke. Previous research suggests that treatments that focus on movement of both hands at the same time or treatments that electrically stimulate the paretic (weak) hand muscles may help the recovery of hand function after stroke. In this study, two electrical stimulation treatments will be compared in their effectiveness in restoring hand movement and hand function. One of the treatments is stimulation only, and the other is stimulation linked to movement of the contralateral hand.

Study participants will be stroke survivors who are enrolled while they are still within their first 6 months after their stroke. After enrolling, their hand movement and function will be tested. Then they will be randomly assigned to one of the two treatments. Each treatment will last 6 weeks. The treatment will require the participant to perform specific exercises at home for a total of 2 hours every day and to come to the laboratory twice a week for study-related occupational therapy. At the end of the 6-week treatment, tests of hand movement and hand function will be repeated. The same tests will be repeated again at 1 and 3 months after the end of treatment to see if the effects of the treatment persist as time goes on. Changes in upper extremity impairment and activity limitation will be compared across treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Within 6 months of first clinical hemorrhagic or nonhemorrhagic stroke
* Cortical or subcortical stroke
* Unilateral upper extremity hemiparesis with severe finger extensor and flexor paresis (<= grade 4 on Medical Research Council (MRC) scale)
* Adequate movement of the shoulder and elbow to allow volitional positioning of the affected hand in the workspace.
* Surface NMES of finger and thumb extensors produces functional hand opening without pain
* Full volitional opening of the contralateral hand of the unimpaired side.
* Able to follow 3 stage commands
* Able to remember at least 2 of 3 items after 30 minutes
* Able to hear and respond (by opening the less affected hand) to auditory cues issued from the stimulator?
* Caregiver available and willing to help assist with the device and home regimen and ensure compliance
* Skin intact on hemiparetic arm
* Medically stable

Exclusion Criteria:

* Insensate forearm and/or hand
* Edema of the affected forearm and/or hand
* History of potentially fatal cardiac arrhythmias.
* Cardiac pacemakers or any other implanted electronic systems
* Pregnant women
* Uncontrolled seizure disorder
* Severely impaired cognition or comprehension
* Uncompensated hemineglect
* Severe depression (>= 13 on Beck Depression Inventory Fast Screen)
* Ipsilateral lower motor neuron lesion
* Parkinson's Disease
* Spinal cord injury
* Traumatic brain injury
* Multiple sclerosis
* Lack of functional passive range of motion of the wrist or fingers of affected side
* Severe shoulder or hand pain (unable to volitionally position hand in the workspace without pain)
* Intramuscular botulinum toxin injections in upper extremity muscle in the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayme S Knutson, PhD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knutson JS, Harley MY, Hisel TZ, Chae J. Improving hand function in stroke survivors: a pilot study of contralaterally controlled functional electric stimulation in chronic hemiplegia. Arch Phys Med Rehabil. 2007 Apr;88(4):513-20. doi: 10.1016/j.apmr.2007.01.003. PMID 17398254
- [Background] Glanz M, Klawansky S, Stason W, Berkey C, Chalmers TC. Functional electrostimulation in poststroke rehabilitation: a meta-analysis of the randomized controlled trials. Arch Phys Med Rehabil. 1996 Jun;77(6):549-53. doi: 10.1016/s0003-9993(96)90293-2. PMID 8831470
- [Background] Chae J, Bethoux F, Bohine T, Dobos L, Davis T, Friedl A. Neuromuscular stimulation for upper extremity motor and functional recovery in acute hemiplegia. Stroke. 1998 May;29(5):975-9. doi: 10.1161/01.str.29.5.975. PMID 9596245
- [Background] Luft AR, McCombe-Waller S, Whitall J, Forrester LW, Macko R, Sorkin JD, Schulz JB, Goldberg AP, Hanley DF. Repetitive bilateral arm training and motor cortex activation in chronic stroke: a randomized controlled trial. JAMA. 2004 Oct 20;292(15):1853-61. doi: 10.1001/jama.292.15.1853. PMID 15494583
- [Background] Whitall J, McCombe Waller S, Silver KH, Macko RF. Repetitive bilateral arm training with rhythmic auditory cueing improves motor function in chronic hemiparetic stroke. Stroke. 2000 Oct;31(10):2390-5. doi: 10.1161/01.str.31.10.2390. PMID 11022069
- [Background] Mudie MH, Matyas TA. Can simultaneous bilateral movement involve the undamaged hemisphere in reconstruction of neural networks damaged by stroke? Disabil Rehabil. 2000 Jan 10-20;22(1-2):23-37. doi: 10.1080/096382800297097. PMID 10661755
- See also: Cleveland FES Center — http://fescenter.org/index.php
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org/body.cfm?id=2438

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CCFES | cNMES
Started | 10 | 11
Completed | 9 | 8
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCFES | cNMES | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.9) | 43.9 (15.2) | 48.6 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Voluntary Finger Extension Angle (a Measure of Hand Impairment)
Description: A custom-built electrogoniometer recorded the angles of the metacarpophalangeal (MP) and proximal interphalangeal (PIP) joints of the index finger simultaneously. Participants were seated with the forearm and wrist supported and stabilized in a neutral posture. From this resting postion, they were instructed to extend their fingers as fully as possible in response to a 4-sec audio cue. The MP and PIP angles were added together, providing a composite measure of degree of finger extension, where 0 degrees corresponds to full extension of the MP and PIP joints. The more negative the angle, the more flexed the finger.
Time Frame: 3 months post-treatment.
Population: The participants who completed the 6-week treatment phase were included in the analysis.
Measure: Mean (Standard Error); unit: degrees
Arm/Group | CCFES | cNMES
Number analyzed (Participants) | 9 | 8
degrees | -11.6 (11.7) | -43.4 (12.5)

2. Secondary Outcome: Finger Tracking Error
Description: A 30-sec 0.1Hz sine wave track scrolled from right to left on a computer screen in front of the participant. The amplitude of the sine wave was scaled to match the middle 70% of the participant's voluntary finger active range of motion (AROM). A cursor on the computer screen moved up and down as the participant extended and flexed their index finger. The task was to trace the scrolling sine wave with the cursor. Tracking error was the average vertical distance between the cursor and the target trace. Since the track was scaled to the participant's finger AROM, the distance between the cursor and the target trace (and therefore the tracking error) is in units corresponding to the percentage (%) of the participant's finger active range of motion (AROM), hereafter abbreviated %AROM.
Time Frame: 3 months post-treatment.
Population: The participants who completed the 6-week treatment phase were included in the analysis.
Measure: Mean (Standard Error); unit: % AROM
Arm/Group | CCFES | cNMES
Number analyzed (Participants) | 9 | 8
% AROM | 4.7 (1.9) | 8.3 (2.0)

3. Secondary Outcome: Box and Blocks Score
Description: The number of blocks picked up and moved across a barrier in 60 seconds
Time Frame: 3 months post-treatment.
Population: The participants who completed the 6-week treatment phase were included in the analysis.
Measure: Mean (Standard Error); unit: blocks
Arm/Group | CCFES | cNMES
Number analyzed (Participants) | 9 | 8
blocks | 29.8 (3.8) | 22.9 (4.1)

4. Secondary Outcome: Arm Motor Abilities Test
Description: The Arm Motor Abilities Test (AMAT) score is an average across 9 different compound activities of daily living (ADL) tasks composed of 1 to 3 component tasks, each of which was scored by a therapist using a 0 to 5 ordinal scale: 0, no attempt to use affected limb; 1, attempt to use affected limb but it doesn't participate functionally; 2, affected limb is used only as a helper or stabilizer; 3, affected limb is used slowly or within synergy patterns; 4, affected limb use almost normal; 5, normal use. Each of the 9 tasks is scored and then the average score across the 9 tasks is calculated, with a range of 0 to 5.
Time Frame: 3 months post-treatment.
Population: The participants who completed the 6-week treatment phase were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CCFES | cNMES
Number analyzed (Participants) | 9 | 8
units on a scale | 3.54 (0.27) | 3.20 (0.29)

5. Secondary Outcome: Fugl-Meyer Assessment (Upper Extremity)
Description: The participant was asked to perform specific coordinated and isolated shoulder, elbow, wrist, and hand movements. Each movement was rated by a therapist using a 3-point ordinal scale: 0, cannot perform; 1, perform partially; 2, perform fully) and summed to produce an overall score, with a range of 0 to 66 (the higher the score the better).
Time Frame: 3 months post-treatment.
Population: The participants who completed the 6-week treatment phase were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CCFES | cNMES
Number analyzed (Participants) | 9 | 8
units on a scale | 46.2 (2.1) | 41.1 (2.2)

ADVERSE EVENTS:
Arm/Group | CCFES | cNMES
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No